CLINICAL TRIAL: NCT02098720
Title: An Open, Non-randomize, Single-center, Safety and Efficacy Study of Conbercept in Patients With Very Low Vision Secondary to Wet Age-related Macular Degeneration
Brief Title: An Open, Single-center, Safety and Efficacy Study of Conbercept in Patients With Very Low Vision Secondary to Wet Age-related Macular Degeneration (wAMD)
Acronym: LAMP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHSWKH902009
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Very Low Vision Secondary to Wet Age-related Macular Degeneration
MeSH Terms: interventions — KH902 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Conbercept (Experimental): Subjects will receive Conbercept injections at a dose of 0.5 mg/eye, once a month for first 3 months. In the next 3 months, the investigator will decide whether repeat injections are needed based on the monthly assessment results.
  Interventions: Drug: Conbercept

INTERVENTIONS:
Drug: Conbercept

SUMMARY:
This study is designed to evaluate the effect of Conbercept therapy on visual acuity and anatomic outcomes and safety observed in subjects with very low vision secondary to wet age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients give fully informed consent and are willing and able to comply with all study procedures.
2. In the study eye:

   There are primary or recurrent subfoveal or parafoveal active choroidal neovascularization (CNV) lesions secondary to wAMD.

   The criterion of active CNV should meet at least one of following three conditions :
   * fresh bleeding;
   * neurosensory detachment showed on optical coherence tomography(OCT);
   * leakage showed on fundus fluorescein angiography (FFA).
3. BCVA in study eye < 19 letters (approximately 20/400 Snellen equivalent).

Exclusion Criteria:

1. Past or existing non-exudative AMD in study eye decided by investigator that have affected macular detection or central vision;
2. Subretinal hemorrhage in study eye and bleeding area ≥6 disc areas;
3. History of vitreous hemorrhage within last month;
4. The maximum diameter of scar and fibrosis area ≥500μm at subfoveal in study eye;
5. Photodynamic therapy (PDT) or drug treatment of CNV within last 6 months in study eye, or anti-vascular endothelial growth factor (VEGF) therapy in fellow eye within last month;
6. History of glaucoma in study eye;
7. Aphakia (excluding artificial lens) in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
percentage of patients with best corrected visual acuity (BCVA ) ≥19 letters gain | 6-month

SECONDARY OUTCOMES:
mean change in BCVA from baseline | 6-month
change from baseline of macular area thickness and other anatomy results | 6-month
safety of Conbercept therapy | 6-month
  To assess incidence of adverse events, incidence of adverse drug reactions etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center,Sun yat-sen University, Guangzhou, Guangdong, China